CLINICAL TRIAL: NCT04363216
Title: Pharmacologic Ascorbic Acid as an Activator of Lymphocyte Signaling for COVID-19 Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JT#15681
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: ascorbic acid; vitamin c
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Ascorbic acid solution (Ascor®, McGuff Pharmaceuticals, Ltd.) will be added to each liter of sterile wate,r plus 1 g/L magnesium chloride to reduce burning sensation, and given parenterally over a 2-hour period. On the day of enrollment (Day 0), 0.3 g/kg will be given; Day 1 - 0.6 g/kg; Day 2 - 0.9 g/kg; Day 3 - 0.9 g/kg; Day 4 - 0.9 g/kg; Day 5 - 0.9 g/kg. After the first dose, each subsequent dose will be given 24 +/- 4 hours following the previous dose.
  Interventions: Drug: Ascorbic Acid
- Routine care (No Intervention): These subject will follow routine care and their clinical courses will be recorded only.

INTERVENTIONS:
Drug: Ascorbic Acid — Ascor® ascorbic acid 2-hour infusion daily (for 6 days), escalating dose (0.3g/kg, 0.6g/kg, 0.9g/kg).
  Other Names: Vitamin C
  Arms: Treatment

SUMMARY:
There are currently no approved therapies for patients with coronavirus disease (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Infusion of ascorbic acid (vitamin C) has been shown to increase activity of lymphocytes, which are a crucial component of the body's defense against viral disease progression and adaptive immunity. Ascorbic acid infusion has been shown to be a safe treatment for patients suffering from sepsis and certain types of cancer. This study is designed to evaluate the safety and efficacy of ascorbic acid in the form of sequential I.V. infusions (Ascor®) for patients with suspected COVID-19 who are unlikely to require mechanical ventilation within 24 hours of study intervention.

DETAILED DESCRIPTION:
Ascorbic acid [AA] (vitamin C) is an essential nutrient that, in addition to aiding tissue repair, also functions as an enzyme co-factor, an antioxidant, and a key component in lymphocyte development and function. Lymphocytes are responsible for adaptive immunity, the immune response following vaccination, in addition to playing a vital role in protection against viral disease progression. Both sepsis and aberrant lymphocyte activation have been associated with severe AA deficiency. We hypothesize that the administration of increasing concentrations of pharmacologic AA promotes lymphocyte activation and signaling in newly admitted, non-ventilator dependent COVID-19 patients via hydrogen peroxide generation and/or DNA de-methylation, and that this will lead to improved clinical outcomes.

This is a single-center, prospective, randomized, open-label, phase II clinical trial designed to assess the efficacy, tolerability, and safety of pharmacologic AA administration in hospitalized patients newly-diagnosed with COVID-19 who will likely not require mechanical ventilation within 24 hours of study intervention. All subjects enrolled will be pending inpatient admission or already admitted as they will require supplemental oxygen. Within 12 hours of admission to the E.D. or medical/surgical floor (rapid screens to determine eligibility must be completed within this time), patients will receive escalating pharmacologic AA over 2 hours once daily for 3 escalating doses, then continued on the highest dose for a total of 6 infusions.

Subjects will be randomized 2:1, with 66 subjects receiving AA treatments and 22 subjects receiving routine clinical care. The open-label design allows investigators to evaluate the safety and clinical progress in real-time. Any subject randomized to AA treatment who is upgraded to ICU-level care, requires high-flow O2 supplementation, or is intubated, will no longer receive AA infusions in order to maximize patient safety during this study. Given the robust safety data on the treatment, a phase II design was chosen with an interim safety analysis after 21 patients. Randomization will be stratified according to high vs. low risk of complications. Patients will be considered to be high risk if they have any of the following characteristics: age>60, hypertension, structural lung disease, cardiovascular disease, diabetes, immunocompromising conditions or meds (such as immunosuppressing meds in transplant patients).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female > 18 years of age at the time of consent
2. ConfirmedSARS-CoV-2 infection
3. Disease severity necessitating hospitalization
4. Currently taking supplemental oxygen
5. No anticipated need (within 24 hours) for mechanical ventilation, defined as:

   1. Positive clinical response to oxygen supplementation with improvement in hypoxia or
   2. Hypoxia improvement with bronchospasm therapy if bronchospasm present

Exclusion Criteria

1. eGFR < 50
2. Known Glucose-6-phosphate dehydrogenase (G6PD) deficiency
3. Anticipated need for mechanical ventilation within 24 hours
4. Pregnant or breastfeeding
5. Requires home oxygen for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | 72 hours
  • Clinical improvement at 72 hours of treatment, defined as a 50% reduction in the highest flow rate of oxygen during the 72 hour period, a 50% reduction in the most frequent use of bronchodilators within a 12-hour window within the 72-hour period, or hospital discharge (whichever comes first).

SECONDARY OUTCOMES:
Patient status upgraded to ICU level [Clinical decline] | 36 hours
  Subject is upgraded to ICU-level care
Oxygen supplementation | up to 1 year
  Overall rate of oxygen supplementation in L/min
Days with fever | up to 1 year
  Number of days during hospitalization where a fever (>100.4°F) is reached at least once
Days to discharge | up to 1 year
  Number of days from initial treatment to hospital discharge
SAEs | up to 1 year
  Serious adverse events specific to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dagan Coppock, M.D., Principal Investigator — Thomas Jefferson University; Daniel Monti, M.D., Study Director — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: No